CLINICAL TRIAL: NCT05044663
Title: Liver and Splenic Stiffness in Predicting Esophageal Varices Needing Treatment in MASLD Related Compensated Advanced Chronic Liver Disease - A Cross-Sectional Study.
Brief Title: Liver and Splenic Stiffness in Predicting Esophageal Varices Needing Treatment in MASLD Related Compensated Advanced Chronic Liver Disease.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-43
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MASLD related cACLD: MASLD related cACLD (Liver Stiffness ≥10 kPa).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Patients with chronic liver disease (CLD) are at risk of developing clinically significant portal hypertension (CSPH). In the Baveno VI consensus a new term "compensated advanced chronic liver disease (cACLD)'' has been proposed to better reflect that the spectrum of severe fibrosis and cirrhosis is a continuum in asymptomatic patients. Liver stiffness by TE is sufficient to suspect cACLD in asymptomatic subjects with known causes of CLD. TE values <10 kPa in the absence of other known clinical signs rule out cACLD; values between 10 and 15 kPa are suggestive of cACLD but need further test for confirmation; values >15 kPa are highly suggestive of cACLD. Patients with a liver stiffness <20 kPa and with a platelet count >150,000 have a < 5 % risk of having varices requiring treatment, and can avoid screening endoscopy. SSM can also predict the presence of CSPH and varices requiring treatment. Because of restrictive nature of Baveno VI, recent Baveno VII guidelines state that patients not satisfying Baveno VI criterai acan have endoscopy avoided if their spleen stiffness is less than 40kPa. Some studies have shown superiority of splenic stiffness over liver stiffness in predicting varices requiring treatment likely attributable to the better performance of SSM compared with LSM in more severe portal hypertension because it reflects better the hemodynamic component of portal hypertension. However, there are few studies on MASLD and most are on viral hepatitis related cACLD. Moreover, very few studies are published on splenic stiffness from Indian subcontinent. Hence, we intend to do the study assessing diagnostic utility of splenic and liver stiffness and validate the Baveno VII algorothm in predicting varices needing treatment in MASLD related cACLD and compare from other noninvasive markers.

ELIGIBILITY:
Inclusion Criteria:

* MASLD will be diagnosed by liver biopsy or ultrasound steatosis / Fibroscan CAP > 250 dB + any 1 criteria of metabolic syndrome:

  1. Waist circumference 90 ≥ cm for males or ≥80 cm for females
  2. Triglycerides ≥150 mg/dL
  3. HDL-C < 40 mg/dL in males or < 50 mg/dl in females
  4. systolic blood pressure (SBP) ≥130 mm Hg or diastolic blood pressure (DBP) ≥ 85 mmHg or both and
  5. Fasting plasma glucose ≥ 100 mg/dL. cACLD is defined with Liver stiffness ≥10 kPa. Ultrasound examination, blood examination and upper gastrointestinal endoscopy will be performed within 1 month of Fibroscan examination. HVPG if indicated will be done within 1 month of Fibroscan.

Exclusion Criteria:

1. Age < 18 and > 70 years, Other etiologies of liver disease.
2. Past or present history of decompensation (ascites, variceal bleed, hepatic encephalopathy, jaundice),
3. Child Pugh B or C,
4. unreliable liver and splenic stiffness in Fibroscan examination,
5. Transjugular intrahepatic portosystemic shunt, significant alcohol intake (> 30 gm/day (M) and 20gm/day (F),
6. Acute on chronic liver failure,
7. AST and/or ALT > 5 times the upper limit of normal.
8. Hepatocellular carcinoma or any space-occupying lesion in the liver,
9. Portal vein thrombosis,
10. Biliary obstruction,
11. HVOTO,
12. Cardiac failure,
13. Prior variceal endotherapy or ongoing beta blocker treatment.
14. HIV,
15. Any malignancy,
16. Pregnancy,
17. ICD / pacemaker,
18. No consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of MASLD related cACLD (Liver Stiffness ≥10 kPa).
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Utility of BAVENO 7 criteria to predict presence of esophageal varices needing treatment in patients of MASLD related cACLD. | Day 0

SECONDARY OUTCOMES:
Utility of other NITs in predicting VNT in MASLD related cACLD | Day 0
Correlation of LSM and SSM with grade of EV | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided